CLINICAL TRIAL: NCT01783704
Title: Improving Community Ambulation After Hip Fracture
Acronym: CAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Arcadia University (Other); UConn Health (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Jay S. Magaziner, Professor and Chair, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HP-00046956; 1R01AG035009-01A1 (NIH)
Record Dates: First submitted 2013-01-31; First posted 2013-02-05 (Estimated); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Hip Fracture
Keywords: hip fracture; randomized controlled trial; exercise
MeSH Terms: conditions — Hip Fractures; Motor Activity | interventions — Nutritional Status; Pulse

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Study PI (Magaziner) and Co-PI (Craik) and members of the Clinical Coordinating Center (Orwig, Lewis) are blinded to treatment assignment.
  Clinical site PIs and clinical site coordinators who are responsible for assigning work and/or assessing for treatment fidelity of PTs in both groups are unblinded.
  Staff who perform evaluations (clinical site visits and telephone interviews) after randomization and the Independent Safety Monitor (ISM) who will be blinded to treatment assignment.
  The PTs only know specific information about the intervention he/she is delivering. To minimize "contamination" of the interventions, each PT provides only one of the interventions and PTs do not have contact with participants in the other group or with PTs providing the intervention to the other group. As PTs are hired for the study, they are assigned at random to one of the interventions.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PUSH and Nutrition (Experimental): PUSH is a specific multi-component intervention based on improving specific precursors to community ambulation. The intervention addresses endurance with continuous upright exercise for 20 min.; function by improving fast walking, standing from a chair, and stair negotiation; muscle performance by exercising to enhance lower extremity strength; and balance by performing unilateral activities and activities with decreased base of support. Participants receive 32 visits of approximately 60 minutes in duration from a study PT. Participants will receive up to three visits a week, on non-consecutive days, for 16 weeks. Visits take place in the participant's place of residence. Participants also receive the nutritional intervention for the duration of the 16-week study.
  Interventions: Dietary Supplement: Nutrition; Behavioral: PUSH
- PULSE and Nutrition (Experimental): PULSE is a non-specific multi-component intervention in which participants will receive flexibility exercises, active range of motion (AROM) for the upper and lower extremities, breathing exercises, and transcutaneous electrical nerve stimulation (TENS). Participants receive 32 visits of approximately 60 minutes in duration from a study PT. Participants will receive up to three visits a week, on non-consecutive days, for 16 weeks. Visits will take place in the participant's place of residence. Participants will also receive the nutritional intervention for the duration of the 16-week study.
  Interventions: Dietary Supplement: Nutrition; Behavioral: PULSE

INTERVENTIONS:
Dietary Supplement: Nutrition — Participants receive 2000 IU vitamin D3, 600 mg calcium, and a multivitamin daily for the duration of the study. Nutritional counseling is also provided. Participants are screened at time of randomization to assess nutritional risk using the Mini Nutritional Assessment-Short Form and contacted by a registered dietician (RD) within 7 days of randomization. Those who score ≤7 (malnourished) and participants with baseline serum albumin 2.5-3.5 g/dl receive a visit from an RD with follow-up a week later. Participants who score 8-11 (at risk of malnutrition) and have serum albumin level >3.5 g/dl receive a phone call from the RD and may receive an in-person visit if warranted. Those screening in the normal range (12-14) and have serum albumin level >3.5 g/dl receive a phone call from the RD. Weight is monitored every 4 weeks. Those who lose 2% or more body weight receive a call from the RD. Those who lose 5% or more body weight between baseline and follow-up may be referred to an RD.
Behavioral: PUSH — Strength components of the muscle performance intervention are performed using a portable progressive resistive exercise device (Shuttle® MiniPress, Contemporary Design Company, P.O. Box 5089, Glacier, Washington 98244). Muscle performance focuses on bilateral hip extensors, hip abductors, knee extensors, and plantar flexors. Balance and strength are addressed with additional exercises performed while standing. The endurance intervention begins with 2-3 minutes of continuous upper and lower extremity active range of motion (AROM) with the participant sitting in order to increase the participants' heart rate (HR) or exertion closer to the target zone. The participant is then asked to walk on level surfaces and/or up and down steps to keep the HR within the training zone for 20 minutes.
  Arms: PUSH and Nutrition
Behavioral: PULSE — During the AROM exercises, participants work to increase flexibility and range of motion. Exercises include the neck, shoulders, arms, trunk, hips, knees and ankles. During all AROM exercises, the participant focuses on deep breathing techniques. The second part of the session uses transcutaneous electrical nerve stimulation (TENS) on lower extremity muscle groups to decrease pain, thereby allowing greater ease of mobility. TENS uses low-level electrical current to stimulate superficial cutaneous nerve fibers through the skin. Flexible carbonized, disposable electrodes coated with a self-adhesive conductive polymer will be applied to the skin bilaterally near the motor points on muscle bellies (the gluteal complex, the quadriceps, and the gastrocnemius) for 7 minutes per muscle group.
  Arms: PULSE and Nutrition

SUMMARY:
Activity and exercise are believed to be of benefit for reducing disability in older adults, yet the majority of older adults do not participate in regular exercise and is not active. This is especially true for older adults following hip fracture after they complete the usual rehabilitation program.

This study is being done to compare two 16-week supervised multi-part physical therapy programs (interventions) initiated up to 26 weeks after hip fracture. The investigators want to test whether the interventions lead to improvements in a person's ability to walk on their own in the home and in the local community. With this knowledge the investigators hope to help a greater number of hip fracture patients enjoy a more complete recovery and improved overall health.

ANCILLARY STUDY #1 - MECHANISTIC PATHWAYS TO COMMUNITY AMBULATION (CAP-MP) The goal of this ancillary study is to investigate several mechanisms thought to be related to recovery in ambulatory ability after hip fracture. Selected mechanistic pathways are being investigated by obtaining mechanistic measurements of the participants randomized in the University of Maryland, Baltimore (UMB) clinical site of CAP.

ANCILLARY STUDY #2 - DIET AND DIETARY PATTERNS IN OLDER ADULTS UNDERGOING HIP FRACTURE REHABILITATION The goal of this ancillary study is to analyze dietary patterns for the nutritional characterization of older adults recovering from a hip fracture. The identified dietary patterns, as well as motivators and barriers to intake, will be assessed for their impact on the rate of return to community ambulation in participants randomized at the University of Connecticut Health Center (UCHC) clinical site of CAP.

ANCILLARY STUDY #3 - ROLE OF GLUCOSE METABOLISM IN STRENGTH AND FUNCTIONAL RECOVERY AFTER HIP FRACTURE The goal of this ancillary study is to assess the impact of glucose metabolism on strength and functional performance following resistance training in participants randomized at the UCHC clinical site of CAP.

ANCILLARY STUDY #4 - MUSCLE MECHANISMS UNDERLYING RECOVERY OF FUNCTION AFTER HIP FRACTURE The goal of this ancillary study is to understand some of the key muscle mechanisms associated with recovery in community ambulation following hip fracture in response to the two interventions for participants randomized at the Arcadia University (AU) clinical site of CAP.

DETAILED DESCRIPTION:
MAIN STUDY

Despite improvements in medical management, significant residual disability remains in older persons after a hip fracture. The goal of current clinical practice is independent, safe household ambulation two to three months after surgery. Hip fracture-acquired dependency in functional activities of daily living persists well beyond three months post-surgery. This residual disability indicates that current standard Medicare-reimbursed post-hip fracture rehabilitation (i.e., usual care) fails to return many patients to pre-fracture levels of function. In contrast to stroke and heart disease, other commonly occurring acute conditions in the older population, there are few intervention trials focused on decreasing disability following hip fracture. None of the trials for hip fracture has examined the effect of early post-fracture intervention on the ability to ambulate at a level required for independent function in the community (i.e., community ambulation). Thus, there is a paucity of evidence to justify extending medical management beyond usual care in persons following hip fracture to achieve community, rather than merely household, ambulation.

A randomized controlled trial (RCT) including 210 older adults who have experienced a hip fracture will be carried out at three clinical sites with half of the subjects receiving a specific multi-component intervention (PUSH) and the other half receiving a non-specific multi-component intervention (PULSE). Randomization of 210 participants meeting eligibility criteria will take place after post-acute rehabilitation ends, approximately 6 months (26 weeks) after admission to the hospital for hip fracture. The primary endpoint will be measured using the Six-Minute Walk Test (SMWT) at the end of the 16-week intervention period. The goal is to enable older adults who have experienced a hip fracture to recover sufficiently to become community ambulators.

Primary Aim The primary aim of the study is to determine if a specific multi-component 16-week intervention based on aerobic conditioning, specificity of training, and muscle overload (the PUSH intervention), initiated within 26 weeks of admission to the hospital for hip fracture, will be more successful in producing community ambulation at 16 weeks after randomization than a non-specific multi-component intervention of transcutaneous electrical nerve stimulation (TENS), flexibility activities, and active range of motion exercises (AROM) (the PULSE intervention).

Secondary Aims

1. To determine whether the proportion of community ambulators differs between the PUSH and PULSE interventions at 40 weeks post-randomization and whether the difference in proportions at 40 weeks changed from the difference in proportions at 16 weeks
2. To compare the PUSH and PULSE interventions at 16 weeks and 40 weeks post-randomization with respect to five secondary outcomes that are thought to be precursors to community ambulation (endurance, dynamic balance, walking speed, quadriceps strength, and lower extremity function)
3. To compare the PUSH and PULSE interventions at 16 weeks and 40 weeks post-randomization with respect to several tertiary outcomes (activities of daily living, quality of life, physical activity, lower extremity physical performance, balance confidence, increase of 50 meters or more in distance walked in six minutes, nutritional status, cognitive status, and depressive symptoms)
4. To compare the economic value of the PUSH and PULSE interventions by estimating the impact of the interventions on cost per quality-adjusted life year (QALY) gained over the follow-up period.

In addition to study outcome measures, expected adverse events (AEs) will be assessed every four weeks during a telephone interview. Information about reportable adverse events (RAEs), which include serious adverse events (SAEs), unexpected AEs, or injury that occurs under supervision by study staff, will be collected throughout the study. Vitamin D, calcium, and multivitamin adherence will be monitored by pill counts every four weeks during the intervention period and by self-report during the 4-week telephone calls. Adherence with the PT interventions will also be monitored.

For participants randomized prior to version 10.0 of the protocol, follow-up assessment visits occurred 16 weeks and 40 weeks from the date of randomization and telephone interviews were conducted every four weeks during the 40-week study period for a total of 10 telephone interviews. For participants consented under version 10.0 of the protocol, all follow-up will end at 16 weeks post-randomization. In version 11.0 of the protocol, we will eliminate several secondary and tertiary outcome measures. In the description of outcome measures, we identify the measures that will not be collected for participants consented under protocol version 11.0 or later.

ANCILLARY STUDIES

ANCILLARY STUDY #1 - MECHANISTIC PATHWAYS TO COMMUNITY AMBULATION (CAP-MP) - Dr. Jay Magaziner [Ancillary Study #1 Start Date: April 12, 2014; Primary Completion Date: October 19, 2017; n=39] The CAP-MP ancillary study is intended to supplement the information gained from the parent CAP study, to help investigators understand how older adults recover after injury. Participants enrolled in the CAP parent study at the Baltimore site are invited to participate in the CAP-MP ancillary study and undergo additional testing at the same time points as for the parent CAP study. The objective of the CAP-MP ancillary study is to examine mechanistic factors hypothesized to be on the pathway between two 16-week interventions post-hip fracture and recovery and the ability to ambulate independently in the community. The effect of the interventions on these factors 24 weeks after the intervention ends also will be evaluated. The outcomes for the CAP-MP ancillary study are secondary or tertiary to the main CAP study.

Primary Aim. To determine if, at the end of the 16-week intervention, participants in the PUSH group, compared to the PULSE group, have: a) greater muscle volume and attenuation (i.e., reduced intra-muscular fat) of the thigh; b) greater lower extremity strength; c) greater bone mineral density and bone strength; d) more bone formation and less bone resorption; e) lower levels of circulating inflammatory cytokines; f) higher levels of the hormones insulin-like growth factor (IGF)-1, testosterone, and estradiol; g) greater aerobic capacity; h) greater improvement in gait and balance; and i) better cognition and fewer depressive symptoms.

Secondary Aim 1. To determine the long-term (i.e., 24 weeks after intervention ends) effect of the intervention on the mechanistic factors detailed in the primary aim.

Secondary Aim 2. To evaluate the relationships between mechanistic factors detailed in the primary aim above and community ambulatory ability at the end of the intervention and 24 weeks later in order to identify those mechanisms that are most responsible for the ability to ambulate in the community following delivery of the intervention.

Tertiary Aim. To quantify the mediating effect of mechanistic factors detailed in the primary aim on the relationship between the intervention and ability to ambulate in the community at the end of the intervention (16 weeks post-randomization) and 24 weeks later.

ANCILLARY STUDY #2 - DIET AND DIETARY PATTERNS IN OLDER ADULTS UNDERGOING HIP FRACTURE REHABILITATION - Dr. Anne Kenny [n=11] This ancillary study will analyze dietary patterns for the nutritional characterization of older adults recovering from a hip fracture. The identified dietary patterns, as well as motivators and barriers to intake, will be assessed for their impact on the rate of return to community ambulation in the CAP study.

Hypothesis: Those who consume dietary patterns similar to a Mediterranean style diet will have less malnutrition with greater likelihood for a return to community ambulation.

Aim 1. At baseline determine degree of Mediterranean style diet intake and dietary patterns in our sample of hip fracture patients to correlate with nutritional status assessed by the Mini Nutritional Assessment tool (MNA).

Aim 2. Determine motivators and barriers to intake in the hip fracture rehabilitation population and associate with dietary patterns and nutritional status.

Aim 3. Diets determined at baseline will be used to predict community ambulation and similar primary endpoints for CAP.

ANCILLARY STUDY #3 - ROLE OF GLUCOSE METABOLISM IN STRENGTH AND FUNCTIONAL RECOVERY AFTER HIP FRACTURE - Dr. Anne Kenny [n=21] The goal of this ancillary study is to assess the impact of glucose metabolism on strength and functional performance following resistance training in the population. Data on rehabilitation capacity post-fracture in those with diabetes mellitus (DM) are limited and mixed. Studies focusing on rehabilitation potential in DM demonstrate either no impact or a decrease in functional recovery.

Hypothesis: Community-dwelling ambulatory hip fracture survivors with impaired glucose metabolism (measured as homeostasis model assessment-estimated insulin resistance [HOMA- IR] or diagnosis of DM) will not recover lower extremity strength or function as well as those with normal glucose metabolism in response to resistance exercise compared to non-resistance training. Further, investigators propose that higher AGE (measured as pentosidine level and its receptor) will impair strength and functional improvement with resistance exercise. Those with IR and DM have lower IGF-1 and higher levels of IGF binding proteins (IGFBP1 and 3) further limiting the available IGF-1 for tissue use. Investigators hypothesize that the strength and functional improvement from resistance exercise will be mitigated by higher IGFBP in those with DM and IR compared to those with normal glucose metabolism.

Aim 1. To compare change in strength and function between those with diabetes mellitus, insulin resistance, or without either condition compared between two multi-component exercise interventions in which one includes resistance.

Aim 2. To determine association between baseline AGE and IGF/IGFBP on strength and functional improvement and evaluate contribution of change in biomarkers to muscle/function response from resistance exercise.

ANCILLARY STUDY #4 - MUSCLE MECHANISMS UNDERLYING RECOVERY OF FUNCTION AFTER HIP FRACTURE - Dr. Marty Eastlack [Ancillary Study #4 Start Date: April 6, 2015; Primary Completion Date: December 13, 2017; n=22] The purpose of this ancillary study is, therefore, to examine the effect of the two interventions on the precursors to participation in the community.

Hypothesis: Those who participate in the PUSH intervention will have less impairment in body structure and function (muscle thickness and echo intensity), fewer limitations in activities (chair rate of rise and fast gait speed) and therefore better likelihood to return to participation (community ambulation).

Aim 1: To determine if there is a difference between PUSH and PULSE with respect to change in muscle quality (muscle thickness and echo intensity), muscle power (chair rate of rise) and fast gait speed.

Aim 2: To see if differences persist 40 weeks post-randomization. Aim 3: To see if changes in muscle quality predict faster gait speed, chair rate of rise and chair rise strategy (this is categorical) among all participants.

Aim 4: To describe the quality of movement (chair rise strategy and capacity, standing symmetry, temporospatial aspects of gait) among all participants.

Aim 5: To confirm that rate of rise in standing is a proxy for instrumented measure of lower extremity power.

ELIGIBILITY:
Inclusion Criteria:

* Closed fracture of proximal femur
* Age 60 or older at time of randomization
* Minimal trauma fracture
* Non-pathologic fracture
* Surgical fixation of fracture
* Living in the community at time of fracture
* Ambulating without human assistance 2 months prior to fracture
* Unable to walk 300 m or more in 6 minutes without human assistance at time of randomization

Exclusion Criteria:

* Not English speaking
* Does not live within reasonable distance of the clinical center
* End stage renal disease on dialysis
* Recent myocardial infarction
* Uncompensated congestive heart failure
* Lower extremity amputation
* Symptoms of angina pectoris
* Chest pain or shortness of breath (including from severe COPD)
* Participant plans to move out of area or otherwise be unavailable during the 16-week intervention period
* Participation in another clinical trial
* Not community-residing (e.g., resident of a skilled nursing facility) at time of randomization
* Not fully weight-bearing on fractured leg or non-fractured leg at time of randomization
* Calculated creatinine clearance < 15 ml/min
* Serum albumin < 2.5 g/dl
* Hemoglobin < 9 g/dl
* Receiving physical therapy for the hip fracture in the hospital or inpatient rehabilitation facility at time of randomization
* Severely diminished lower extremity sensation or ulceration
* Uncontrolled hypertension
* Denied medical clearance by appropriate medical provider
* Clinical site clinician thinks participant is not a good candidate for study (e.g., not likely to survive study period)
* Cognitive impairment (3MS score <73)
* Development of chest pain or substantial shortness of breath or ambulating with severe pain during baseline SMWT
* Participant walks less than 4 meters in 40 seconds (<0.1 m/sec) during baseline SMWT
* Not randomized by 26 weeks post admission for hip fracture
* Final sign-off from study clinician and/or principal investigator is incomplete
* Incomplete baseline data
* Unable to contact participant
* Participant is unable to provide her/his own informed consent
* Participant refuses the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-06-10 (Actual); Primary Completion 2017-10-17 (Actual); Study Completion 2017-10-17 (Actual)

PRIMARY OUTCOMES:
Ability to walk 300 meters or more in six minutes | 16 weeks post-randomization
  The primary study outcome reflects the concept of a minimum distance a person needs to be able to walk to carry out usual activities in the community. This will be defined as achieving the threshold value of 300 meters or more on the Six-Minute Walk Test (SMWT). The SMWT is an assessment with excellent psychometric properties, and there is sound justification for a 300 m distance threshold on the SMWT (equivalent to walking at 0.8 m/s) to serve as an indicator for community ambulatory ability.

SECONDARY OUTCOMES:
Ability to walk 300 meters or more in six minutes | 40 weeks post-randomization
  Performance of the SMWT (described above) will be used to determine whether the proportion of community ambulators differs between the PUSH and PULSE interventions at 40 weeks post-randomization and whether the difference in proportions at 40 weeks changed from the difference in proportions at 16 weeks.
Endurance | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  To assess endurance, the SMWT (described above) will be used to obtain a continuous measure of total distance walked in six minutes. The SMWT is highly correlated with workloads, heart rate, oxygen saturation, and dyspnea responses when compared to bicycle ergometry and treadmill exercise tests in older persons. It has been performed by elderly, frail and severely compromised participants who cannot perform standard maximal treadmill or cycle ergometry exercise tests.
Balance | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  We will use an enhanced balance measure that includes the balance subscale of the Short Physical Performance Battery (SPPB) and two additional single leg stands (eyes open and eyes closed), as used in the National Health and Aging Trends Study (NHATS). For the test of standing balance, participants are asked to maintain balance in three positions, characterized by a progressive narrowing of the base support (side-by-side, semi-tandem, and tandem). For each of the three positions, participants are timed to a maximum of 10 seconds. Participants are then asked to stand on one leg (on the side of the fracture) with eyes open and again with eyes closed. Each of the single leg stands are held for up to 30 seconds. The number of seconds is then summed across the 5 items to obtain the measure of balance. These tests are hierarchical such that when a participant fails an item, the harder ones are not administered and receive a score of 0.
Quadriceps muscle strength | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Isometric force for bilateral knee extensors will be measured with a portable, hand-held dynamometer (Microfet2 Manual Muscle Tester). Participants will be seated on the strength testing chair to increase stabilization, with hip flexion 90° and knee flexed to 70°, stabilization straps on the pelvis and thigh, and resistance applied just proximal to the ankle on the anterior surface of the leg. Participants will be asked to push as hard and as fast as possible for five seconds. Three maximal effort trials, with a one-minute rest between trials, will be performed. The reported test-retest reliability with hand-held dynamometry is excellent (r>.90) if tested in one session and in subjects with muscle weakness (intraclass correlation coefficient ≥ .90). The peak force will be recorded for each of the three trials and the highest value will be used.
  This measure will not be collected for participants consented under protocol version 11.0 or later.
Lower extremity function | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  A modified version of the Physical Performance Test (mPPT) will be used to measure lower extremity function at baseline and follow-up. The modification, used by Binder et al., substitutes a chair-rise task and a balance task for writing and eating tasks, in order to emphasize lower extremity function. The modified PPT includes nine standardized tasks that will be timed (e.g., picking up a penny from the floor, standing up five times from a 16-inch chair). The tasks are performed twice and the times from the two trials are averaged. The score for each item ranges from 0 to 4, with 36 representing a perfect score. Test-retest reliability for the modified PPT score is 0.96. Because there is some overlap between the mPPT and SPPB items, we have integrated the two scales so that participant burden is minimized but it is still possible to obtain scores on each of the scales.
Fast walking speed | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Within the mPPT, participants are asked to walk a distance of 50 feet walking quickly but safely. The time required to walk 50 ft will be the measure of fast walking speed.
Cost effectiveness: health care utilization | Every four weeks, up to 16 weeks post-randomization and up to 40 weeks post-randomization for a subset of participants
  The economic value of the interventions will be determined by assessing the impact on quality-adjusted life years (QALYs), cost, and cost per QALY gained over the 16 weeks following randomization. The cost-effectiveness analyses will address both the within trial comparison of the study interventions and a model-based comparison of the study interventions and usual care.
  This measure will not be collected for participants consented under protocol version 11.0 or later.
Short Physical Performance Battery (SPPB) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  The SPPB evaluates lower extremity performance in older persons based on timed short distance walk, repeated chair stands, and a set of balance tests. Each of the tasks is assigned a score ranging from 0 to 4, with 4 indicating the highest level of performance and 0 an inability to complete the test. The test takes about 10-15 minutes to administer and was designed to be administered by a lay interviewer in a setting with limited space. The battery has an excellent safety record. It has been administered to well over 10,000 persons in various studies and no serious injuries are known to have occurred. The SPPB components and total score are derived from normative values obtained from a population-based study.

OTHER OUTCOMES:
Activities of daily living (ADLs) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  We will measure ADLs using the Pepper Assessment Tool for Disability (PAT-D) with two modifications. First, two items (walking a quarter mile and walking across a small room) were added to address perceived gaps in the original PAT-D scale. This modification is consistent with the version used in the Lifestyle Interventions and Independence for Elders study. Second, two items (walking several blocks and lifting heavy objects) were deleted to avoid duplication with other items in the scale. The resulting 19-item scale allows examination of three subscales (basic ADL, functional limitations, and instrumental ADL).
  This measure will not be collected for participants consented under protocol version 11.0 or later.
Quality of life (SF-36) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  We will use an interviewer-administered version of the SF-36, a health survey that assesses quality of life in eight subscales (physical function, social function, role-physical, role-emotional, bodily pain, mental health, general health, and vitality). The measure has been validated as a generic measure of quality of life in many different populations, including patient and non-patient samples.
  This measure will not be collected for participants consented under protocol version 11.0 or later.
Balance confidence | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  The Activities-specific Balance Confidence (ABC) scale is a 16-item measure that asks respondents to rate their confidence in maintaining their balance while doing daily activities. Test-retest reliability, internal consistency, and concurrent validity with fall and physical activity are high. This measure has been used successfully in hip fracture patients.
  This measure will not be collected for participants consented under protocol version 11.0 or later.
Yale Physical Activity Survey (YPAS) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  This interviewer-administered questionnaire includes five categories of common activities related to work, exercise, and recreation performed during a typical week in the past month. The YPAS increases the sensitivity of other physical activity surveys by describing a wider range of lower intensity activities that older adults often engage in. Participation in each activity (hrs/week) will be multiplied by an intensity code (kcal/min) and then summed over all activities to calculate a weekly energy expenditure summary. The measure has been validated against several physiological variables of habitual activity. The YPAS has been used to estimate change in older adults in an exercise intervention program.
  This measure will not be collected for participants consented under protocol version 11.0 or later.
Improvement in walking | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Whether or not there was an increase of at least 50 meters in the distance walked on the SMWT will be assessed as a tertiary outcome. This distance has been shown to be clinically meaningful.
Depressive symptoms | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Depressive symptoms will be measured using the 20-item Center for Epidemiologic Studies Depression (CES-D) scale, which asks about depressive symptoms experienced in the previous week. There is evidence that recovery post-fracture is delayed in the presence of depression. This scale ranges from 0-60 with higher scores indicating greater depression.
Cognitive status | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Cognitive status will be assessed at follow-up using the 3MS.
  This measure will not be collected for participants consented under protocol version 11.0 or later.
Nutritional status | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Nutritional status will be assessed using the Mini Nutritional Assessment-Short Form (MNA®-SF), a validated and widely used malnutrition screening tool. We are using a modified version of the MNA®, approved by the scale's developer (the Nestlé company), to facilitate use as an interviewer-administered tool in a research setting. Scores range from 0 to 14; participants scoring ≤7 will be considered malnourished; those scoring 8-11 will be considered to be at risk of malnutrition; and those scoring 12-14 will be considered to have normal nutritional status.
  This measure will not be collected at follow-up for participants consented under protocol version 12.0 or later.
Ancillary Study #1 - Muscle and fat mass | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Muscle and lean mass will be estimated using dual-energy x-ray absorptiometry (DXA) (GE LUNAR, Madison, WI). DXA calculates fat mass (g) and muscle mass (g) from the total body scan and values are provided in the report produced by the DXA machine. The coefficient of variation of these measurements in our previous studies for fat and lean mass was 1.4% and 1.3%, respectively.
Ancillary Study #1 - Muscle composition: Intramuscular fat and muscle volume | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Intramuscular fat and muscle volume are calculated when analyzing the thigh CT scan. Thigh CT will be performed every 4 cm starting at the patella and ending at the femoral head (Siemens Somatom Sensation 64 Scanner) to quantify skeletal muscle area, total fat area, low density lean tissue area, and muscle attenuation of the thigh. Scans will be analyzed using MIPAV (Medical Image Processing, Analysis and Visualization, v.7.0, NIH). The cross-sectional area of each axial slice will be multiplied by the distance between slices (4 cm) and summed across slices representing volume expressed in cm3. The average attenuation of muscle tissue and the percentage of low-density lean muscle to total muscle volume is associated with skeletal muscle lipid (fat) content, and a measure of muscle quality.
Ancillary Study #1 - Strength | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  A Biodex System 3 PRO dynamometer will measure concentric isokinetic peak normalized joint torque over the entire range of motion (strength) for bilateral ankle plantarflexion-dorsiflexion and knee flexion-extension. Strength is measured in Newton-meters (Nm). Testing will utilize standardized positioning and joint motion excursions. Subjects will perform two blocks of three repetitions with a rest period between blocks.
Ancillary Study #1 - Power | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  A Biodex System 3 PRO dynamometer will measure strength per unit of time (power) for bilateral ankle plantarflexion-dorsiflexion and knee flexion-extension. Power is measured in Watts (W). Testing will utilize standardized positioning and joint motion excursions. Subjects will perform two blocks of three repetitions with a rest period between blocks.
Ancillary Study #1 - Bone mineral density (BMD) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  BMD will be estimated using DXA as described above. DXA of the contralateral (non-fractured) femur will be measured to yield measures of total hip and femoral neck BMD.
Ancillary Study #1 - Bone geometry | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Bone geometry will be measured with the Hip Structural Analysis (HSA) program. The program uses DXA images to derive cross-section dimensions at defined regions traversing the femur, i.e., narrow neck, intertrochanter, and proximal shaft. At each region, BMD, bone cross-sectional area (CSA), outer diameter, cross-sectional moment of inertia, section modulus, and centroid are measured. Estimates of average cortical thickness and buckling ratio are derived using assumptions of cross-section shape.
Ancillary Study #1 - Bone turnover markers | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Bone turnover markers. a) bone formation (serum aminoterminal propeptide of type 1 procollagen; P1NP) and b) bone resorption (serum cross-linked C-telopeptides of type I collagen; CTx-I) will be assessed.
Ancillary Study #1 - Hormones | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  a) Total testosterone (T) will be measured using the liquid chromatography-tandem mass spectrometry (LCMS/MS) method. b) Estradiol (E2) (Ultra-sensitive E2) will be measured by ELISA. c) Insulin-like growth factor-1(IGF-1) will be measured by RIA, using acid ethanol extraction. d) SHBG will be measured by IRMA. e) 25-hydroxyvitamin D (25-OH D) will be measured by RIA using kits supplied by DiaSorin (Stillwater, MN). This assay detects both the D2 and D3, f) Parathyroid hormone, intact (iPTH) will be measured by ELISA.
Ancillary Study #1 - Inflammatory cytokines | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  a) interleukin-6 (IL-6), b) soluble TNF- α receptor 1 (sTNF- αR1), c) IL-1 receptor antagonist (IL-1ra), and d) interleukin-10 (IL-10). All cytokines will me measured in serum by ELISA (R&D Systems Inc., Minneapolis, MN).
Ancillary Study #1 - Aerobic capacity | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  VO2 peak will be measured using a treadmill with a custom constant velocity protocol with open circuit spirometry for measurement of aerobic capacity (Ametek-Thermox) O2 and CO2 analyzers (Sensormedics 2900 metabolic cart with re-breathing cardiac output option) using a method that has been previously employed in subjects with hemiparetic stroke recent hip fracture.
Ancillary Study #1 - Gait and balance (GAITrite) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  A GAITrite instrumented walkway system will measure spatial and temporal gait parameters. Subjects will walk at their safest fast and natural speeds. In addition, the Dynamic Gait Index, a clinical assessment of balance and mobility while walking, will be administered. Measures will include: step length, walking speed, single and double leg support time, and cadence.
Ancillary Study #1 - Gait and balance (Stepping Test) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  Subjects will stand on two separate force platforms with reflective motion detection markers placed on each foot to record stepping kinematics. Visually cued simple and choice stepping reaction time (RT) tasks will evaluate the rapid initiation of forward stepping. Measures will be response, weight transfer, and movement times, number of false starts and stepping performance. Neuromotor and biomechanical features of balance and gait control will be extracted.
Ancillary Study #1 - Gait and balance (Four Square Step Test) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  It was developed as an easily portable and reliably scored test of balance and ambulatory coordination, and standardized locally according to detailed usage in the literature. Essentially, the subject is timed while stepping into "4 squares" over lines or canes placed on the floor in a "+" pattern moving both clockwise then back counter-clockwise. This will be performed by an exercise physiologist or nurse experienced in its application, using an SOP that has been reviewed by PTRS faculty. The rationale for including this test in addition to the more mechanistic gait and stepping tests above includes its well established clinical relevance and ease of interpretation of change in score over time.
Ancillary Study #1 - Cognitive function (Trail Making Test (Trails A & B)) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  The Trail Making Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test can provide information about visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. It is sensitive to detecting cognitive impairment associated with dementia.
Ancillary Study #1 - Cognitive function (Hooper Visual Organization Test (VOT)) | 16 weeks post-randomization and 40 weeks post-randomization for a subset of participants
  The Hooper VOT is a neuropsychological test of visual spatial ability that presents participants with a line drawing of a common object that has been broken into fragments, and asks participants to name what the object would be if reassembled.
Ancillary Study #2 - Food Frequency Questionnaire (FFQ) | Baseline
  Data collected from the Harvard FFQ includes foods, food groups, and frequency of intake that is averaged by respondents to represent intake over the previous year. This questionnaire is validated against diet record for correlations between nutrients and food intake. Participants will complete the FFQ at home, on their own time. Instructions for completion will be altered to report intake since their hip fracture.
Ancillary Study #2 - 24 Hour Dietary Recall | Baseline
  The diet record (DR) provides a snapshot of current intake. The 7-day weighted DR is considered the gold standard for subjective dietary assessment and the 24 hour DR has been validated in older adults. Participants will record all foods and beverages eaten, the amount consumed and time of consumption in the previous 24 hours. Food models, scales, and examples will be provided to guide the participant to most accurately report intake. Participants will be asked if the 24 hour DR is representative of their intake prior to hip fracture.
Ancillary Study #2 - Food Barriers and Motivators Survey | Baseline
  To assess potential reasons for poor intake or post-hip fracture alterations in their eating behaviors, investigators will inquire about barriers and motivators of food intake including: food security, appetite and sensory appeal, oral health, perception of health and resources, and social factors. To meet the needs of this study, investigators will modify other validated surveys. Surveys used in the development of this survey include the Guide to Measuring Household Food Security from the USDA to assess food security; the Simplified Nutritional Appetite Questionnaire (SNAQ) to access appetite; Vailas' Food Enjoyment Questionnaire to identify barriers of intake; and the Food Choice Questionnaire (FCQ) to assess motivators of food intake.
Ancillary Study #4 - Muscle thickness and quality | Baseline, 16 weeks post-randomization, and 40 weeks post-randomization for a subset of participants
  There are no additional exclusion criteria for the ultrasound measures and no known risks associated with these measures as ultrasound does not use ionizing radiation to acquire images. Muscle quality (thickness and echo intensity) of the gluteus medius, rectus femoris, and lateral heads of the gastrocnemius will be measured using an ultrasound unit (GE - LOGIQ e). Participants will be in a private room and asked to lie in side-lying with their hip and lower leg exposed in order to measure the gluteus medius and lateral gastrocnemius. They will be draped with a sheet for modesty as necessary. Participants will then be asked to roll onto their backs with their front thigh exposed in order to measure the rectus femoris. Ultrasonographic images will be taken bilaterally. The images (which have no identifiers; only their study code) will be downloaded onto a computer and later analyzed using Image J.
Ancillary Study #4 - Sit-to-stand (video and forceplate) | Baseline, 16 weeks post-randomization, and 40 weeks post-randomization for a subset of participants
  Participants will do the sit-to-stand (STS) test from both a standard and adjustable height chair (adjusted to 80% of tibial length with shoes). Participants are instructed to place their arms across their chest throughout the STS maneuver. If unable to do this participants are allowed to use their arms. Participants' feet are placed parallel with each foot on a different forceplate with knees at a 90 degree angle; the width is unrestrained, but consistent throughout trials. The STS test includes 3 trials at the participant's preferred speed then 3 trials as fast as and as slow as possible with rest as needed. A video camera is positioned in the frontal and sagittal plane to record the strategy used to rise from the chair. Participants will come to standing onto forceplates that measure vertical ground reaction force under each leg, the rate at which they rise from the chair at three different speed commands, and the time range between fast and slow trials as a measure of capacity.
Ancillary Study #4 - Lower extremity power (Primus) | Baseline, 16 weeks post-randomization, and 40 weeks post-randomization for a subset of participants
  The participant will be placed on a machine (Primus) that will allow the measurement of lower extremity power during the "leg press exercise" movement. First, the participant will be given several practice trials and the test will only begin after they demonstrate understanding of the task. The participant will then be asked to do this movement against three different resistances (set to 30, 40, and 50% of body weight) for a total of up to 15 trials; 5 at each percentage of body weight. We will be looking for 3 trials that are consistent (≤ 5% coefficient of variation among trials) and as soon as this is done the participant will proceed to the next resistance level. In our pilot study with healthy elders (age range 58-88; 75 + 12 yrs) all participants were able to achieve 3 consistent trials within the specified five trials with no adverse events.
Ancillary Study #4 - Temporospatial measures of walking (Gait Mat) | Baseline, 16 weeks post-randomization, and 40 weeks post-randomization for a subset of participants
  Temporal and spatial characteristics of gait will be measured with the Gait Mat II (EQ, Inc., Telford, PA). The participant will be instructed to walk at usual, fast and as slowly as possible without stopping. Individually determined rest periods will be given between the trials. The Gait Mat II ™ is connected to a personal computer and collects average walking speed (m/sec) and calculates step length as the spatial distance between the location of the first switch closure of one footprint and the location of the first switch closure of the previous footprint on the contralateral side. Single support time is calculated as the time from the last switch opening of one step to the first switch closure of the next step. Left single support time is the same as right swing time.

CONTACTS AND LOCATIONS:
Overall Officials: Jay Magaziner, PhD, MSHyg, Study Chair — University of Maryland
Locations (4):
- United States (4):
  - University of Connecticut Health Center, Farmington, Connecticut
  - University of Maryland, Baltimore, Baltimore, Maryland
  - Dartmouth Medical School, Lebanon, New Hampshire
  - Arcadia University, Glenside, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Magaziner J, Fredman L, Hawkes W, Hebel JR, Zimmerman S, Orwig DL, Wehren L. Changes in functional status attributable to hip fracture: a comparison of hip fracture patients to community-dwelling aged. Am J Epidemiol. 2003 Jun 1;157(11):1023-31. doi: 10.1093/aje/kwg081. PMID 12777366
- [Background] Magaziner J, Hawkes W, Hebel JR, Zimmerman SI, Fox KM, Dolan M, Felsenthal G, Kenzora J. Recovery from hip fracture in eight areas of function. J Gerontol A Biol Sci Med Sci. 2000 Sep;55(9):M498-507. doi: 10.1093/gerona/55.9.m498. PMID 10995047
- [Background] Chang KP, Center JR, Nguyen TV, Eisman JA. Incidence of hip and other osteoporotic fractures in elderly men and women: Dubbo Osteoporosis Epidemiology Study. J Bone Miner Res. 2004 Apr;19(4):532-6. doi: 10.1359/JBMR.040109. Epub 2004 Jan 5. PMID 15005838
- [Background] Koval KJ, Cooley MR. Clinical pathway after hip fracture. Disabil Rehabil. 2005 Sep 30-Oct 15;27(18-19):1053-60. doi: 10.1080/09638280500056618. PMID 16278174
- [Background] Enright PL, Sherrill DL. Reference equations for the six-minute walk in healthy adults. Am J Respir Crit Care Med. 1998 Nov;158(5 Pt 1):1384-7. doi: 10.1164/ajrccm.158.5.9710086. PMID 9817683
- [Background] Guyatt GH, Sullivan MJ, Thompson PJ, Fallen EL, Pugsley SO, Taylor DW, Berman LB. The 6-minute walk: a new measure of exercise capacity in patients with chronic heart failure. Can Med Assoc J. 1985 Apr 15;132(8):919-23. PMID 3978515
- [Background] Peeters P, Mets T. The 6-minute walk as an appropriate exercise test in elderly patients with chronic heart failure. J Gerontol A Biol Sci Med Sci. 1996 Jul;51(4):M147-51. doi: 10.1093/gerona/51a.4.m147. PMID 8680996
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] VanSwearingen JM, Brach JS. Making geriatric assessment work: selecting useful measures. Phys Ther. 2001 Jun;81(6):1233-52. PMID 11380279
- [Background] Enright PL, McBurnie MA, Bittner V, Tracy RP, McNamara R, Arnold A, Newman AB; Cardiovascular Health Study. The 6-min walk test: a quick measure of functional status in elderly adults. Chest. 2003 Feb;123(2):387-98. doi: 10.1378/chest.123.2.387. PMID 12576356
- [Background] Freedman VA. Adopting the ICF language for studying late-life disability: a field of dreams? J Gerontol A Biol Sci Med Sci. 2009 Nov;64(11):1172-4; discussion 1175-6. doi: 10.1093/gerona/glp095. Epub 2009 Jul 17. No abstract available. PMID 19617529
- [Background] Bohannon RW. Test-retest reliability of hand-held dynamometry during a single session of strength assessment. Phys Ther. 1986 Feb;66(2):206-9. doi: 10.1093/ptj/66.2.206. PMID 3945674
- [Background] Andrews AW, Thomas MW, Bohannon RW. Normative values for isometric muscle force measurements obtained with hand-held dynamometers. Phys Ther. 1996 Mar;76(3):248-59. doi: 10.1093/ptj/76.3.248. PMID 8602410
- [Background] Bohannon RW. Reference values for extremity muscle strength obtained by hand-held dynamometry from adults aged 20 to 79 years. Arch Phys Med Rehabil. 1997 Jan;78(1):26-32. doi: 10.1016/s0003-9993(97)90005-8. PMID 9014953
- [Background] Bohannon RW, Andrews AW. Interrater reliability of hand-held dynamometry. Phys Ther. 1987 Jun;67(6):931-3. doi: 10.1093/ptj/67.6.931. PMID 3588679
- [Background] Reuben DB, Siu AL. An objective measure of physical function of elderly outpatients. The Physical Performance Test. J Am Geriatr Soc. 1990 Oct;38(10):1105-12. doi: 10.1111/j.1532-5415.1990.tb01373.x. PMID 2229864
- [Background] Binder EF, Brown M, Sinacore DR, Steger-May K, Yarasheski KE, Schechtman KB. Effects of extended outpatient rehabilitation after hip fracture: a randomized controlled trial. JAMA. 2004 Aug 18;292(7):837-46. doi: 10.1001/jama.292.7.837. PMID 15315998
- [Background] Binder EF, Schechtman KB, Ehsani AA, Steger-May K, Brown M, Sinacore DR, Yarasheski KE, Holloszy JO. Effects of exercise training on frailty in community-dwelling older adults: results of a randomized, controlled trial. J Am Geriatr Soc. 2002 Dec;50(12):1921-8. doi: 10.1046/j.1532-5415.2002.50601.x. PMID 12473001
- [Background] Rejeski WJ, Ettinger WH Jr, Schumaker S, James P, Burns R, Elam JT. Assessing performance-related disability in patients with knee osteoarthritis. Osteoarthritis Cartilage. 1995 Sep;3(3):157-67. doi: 10.1016/s1063-4584(05)80050-0. PMID 8581745
- [Background] Rejeski WJ, Ip EH, Marsh AP, Miller ME, Farmer DF. Measuring disability in older adults: the International Classification System of Functioning, Disability and Health (ICF) framework. Geriatr Gerontol Int. 2008 Mar;8(1):48-54. doi: 10.1111/j.1447-0594.2008.00446.x. PMID 18713189
- [Background] Rejeski WJ, Fielding RA, Blair SN, Guralnik JM, Gill TM, Hadley EC, King AC, Kritchevsky SB, Miller ME, Newman AB, Pahor M. The lifestyle interventions and independence for elders (LIFE) pilot study: design and methods. Contemp Clin Trials. 2005 Apr;26(2):141-54. doi: 10.1016/j.cct.2004.12.005. PMID 15837437
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Ware JE, Snow KK, Kosinski M, Gandek B. SF-36 Health Survey: Manual and Interpretation Guide. Boston, Mass.: Nimrod Press; 1993.
- [Background] Lotz JC, Cheal EJ, Hayes WC. Stress distributions within the proximal femur during gait and falls: implications for osteoporotic fracture. Osteoporos Int. 1995;5(4):252-61. doi: 10.1007/BF01774015. PMID 7492864
- [Background] Powell LE, Myers AM. The Activities-specific Balance Confidence (ABC) Scale. J Gerontol A Biol Sci Med Sci. 1995 Jan;50A(1):M28-34. doi: 10.1093/gerona/50a.1.m28. PMID 7814786
- [Background] Hatch J, Gill-Body KM, Portney LG. Determinants of balance confidence in community-dwelling elderly people. Phys Ther. 2003 Dec;83(12):1072-9. PMID 14640866
- [Background] Whitehead C, Miller M, Crotty M. Falls in community-dwelling older persons followinig hip fracture: impact on self-efficacy, balance and handicap. Clin Rehabil. 2003 Dec;17(8):899-906. doi: 10.1191/0269215503cr695oa. PMID 14682563
- [Background] Petrella RJ, Payne M, Myers A, Overend T, Chesworth B. Physical function and fear of falling after hip fracture rehabilitation in the elderly. Am J Phys Med Rehabil. 2000 Mar-Apr;79(2):154-60. doi: 10.1097/00002060-200003000-00008. PMID 10744190
- [Background] Dipietro L, Caspersen CJ, Ostfeld AM, Nadel ER. A survey for assessing physical activity among older adults. Med Sci Sports Exerc. 1993 May;25(5):628-42. PMID 8492692
- [Background] Pescatello L, DiPietro L, Fargo A, Ostfeld A, Nadel E. The impact of physical activity and physical fitness on health indicators among older adults. Journal of Aging and Physical Activity 2: 2-13, 1994.
- [Background] Resnick B, Magaziner J, Orwig D, Zimmerman S. Evaluating the components of the Exercise Plus Program: rationale, theory and implementation. Health Educ Res. 2002 Oct;17(5):648-58. doi: 10.1093/her/17.5.648. PMID 12408209
- [Background] Perera S, Mody SH, Woodman RC, Studenski SA. Meaningful change and responsiveness in common physical performance measures in older adults. J Am Geriatr Soc. 2006 May;54(5):743-9. doi: 10.1111/j.1532-5415.2006.00701.x. PMID 16696738
- [Background] Guralnik JM, Simonsick EM, Ferrucci L, Glynn RJ, Berkman LF, Blazer DG, Scherr PA, Wallace RB. A short physical performance battery assessing lower extremity function: association with self-reported disability and prediction of mortality and nursing home admission. J Gerontol. 1994 Mar;49(2):M85-94. doi: 10.1093/geronj/49.2.m85. PMID 8126356
- [Background] Guralnik JM, Seeman TE, Tinetti ME, Nevitt MC, Berkman LF. Validation and use of performance measures of functioning in a non-disabled older population: MacArthur studies of successful aging. Aging (Milano). 1994 Dec;6(6):410-9. doi: 10.1007/BF03324272. PMID 7748914
- [Background] Guralnik JM, Ferrucci L, Pieper CF, Leveille SG, Markides KS, Ostir GV, Studenski S, Berkman LF, Wallace RB. Lower extremity function and subsequent disability: consistency across studies, predictive models, and value of gait speed alone compared with the short physical performance battery. J Gerontol A Biol Sci Med Sci. 2000 Apr;55(4):M221-31. doi: 10.1093/gerona/55.4.m221. PMID 10811152
- [Background] Radloff LS. The CES-D Scale: A self-report depression scale for research in the general population. Applied psychological measurement 1: 385-401, 1977.
- [Background] Mossey JM, Knott K, Craik R. The effects of persistent depressive symptoms on hip fracture recovery. J Gerontol. 1990 Sep;45(5):M163-8. doi: 10.1093/geronj/45.5.m163. PMID 2394912
- [Background] Zimmerman SI, Smith HD, Gruber-Baldini A, et al. Short-term persistent depression following hip fracture: a risk factor and target to increase resilience in elderly people. Social Work Research 23:187-96, 1999.
- [Background] Sayetta RB, Johnson DP. Basic data on depressive symptomatology. United States, 1974-75. Vital Health Stat 11. 1980 Apr;(216):i-v, 1-37. doi: 10.1037/e531192008-001. No abstract available. PMID 7385607
- [Background] Weissman MM, Sholomskas D, Pottenger M, Prusoff BA, Locke BZ. Assessing depressive symptoms in five psychiatric populations: a validation study. Am J Epidemiol. 1977 Sep;106(3):203-14. doi: 10.1093/oxfordjournals.aje.a112455. PMID 900119
- [Background] Guigoz Y, Vellas B, Garry PJ. Assessing the nutritional status of the elderly: The Mini Nutritional Assessment as part of the geriatric evaluation. Nutr Rev. 1996 Jan;54(1 Pt 2):S59-65. doi: 10.1111/j.1753-4887.1996.tb03793.x. No abstract available. PMID 8919685
- [Background] Kaiser MJ, Bauer JM, Ramsch C, Uter W, Guigoz Y, Cederholm T, Thomas DR, Anthony P, Charlton KE, Maggio M, Tsai AC, Grathwohl D, Vellas B, Sieber CC; MNA-International Group. Validation of the Mini Nutritional Assessment short-form (MNA-SF): a practical tool for identification of nutritional status. J Nutr Health Aging. 2009 Nov;13(9):782-8. doi: 10.1007/s12603-009-0214-7. PMID 19812868
- [Background] Wells JL, Dumbrell AC. Nutrition and aging: assessment and treatment of compromised nutritional status in frail elderly patients. Clin Interv Aging. 2006;1(1):67-79. doi: 10.2147/ciia.2006.1.1.67. PMID 18047259
- [Background] Vellas B, Guigoz Y, Garry PJ, Nourhashemi F, Bennahum D, Lauque S, Albarede JL. The Mini Nutritional Assessment (MNA) and its use in grading the nutritional state of elderly patients. Nutrition. 1999 Feb;15(2):116-22. doi: 10.1016/s0899-9007(98)00171-3. PMID 9990575
- [Background] Rubenstein LZ, Harker JO, Salva A, Guigoz Y, Vellas B. Screening for undernutrition in geriatric practice: developing the short-form mini-nutritional assessment (MNA-SF). J Gerontol A Biol Sci Med Sci. 2001 Jun;56(6):M366-72. doi: 10.1093/gerona/56.6.m366. PMID 11382797
- [Background] Wilson MM, Thomas DR, Rubenstein LZ, Chibnall JT, Anderson S, Baxi A, Diebold MR, Morley JE. Appetite assessment: simple appetite questionnaire predicts weight loss in community-dwelling adults and nursing home residents. Am J Clin Nutr. 2005 Nov;82(5):1074-81. doi: 10.1093/ajcn/82.5.1074. PMID 16280441
- [Background] Bickel G, Nord M, Price C, Hamilton W, Cook J. Guide to Measuring Household Food Security, Revised 2000. In: U.S. Department of Agriculture FaNS, editor. Alexandria, VA 2000.
- [Background] Vailas LI, Nitzke SA, Becker M, Gast J. Risk indicators for malnutrition are associated inversely with quality of life for participants in meal programs for older adults. J Am Diet Assoc. 1998 May;98(5):548-53. doi: 10.1016/S0002-8223(98)00123-0. PMID 9597027
- [Background] Locher JL, Ritchie CS, Roth DL, Sen B, Vickers KS, Vailas LI. Food choice among homebound older adults: motivations and perceived barriers. J Nutr Health Aging. 2009 Oct;13(8):659-64. doi: 10.1007/s12603-009-0194-7. PMID 19657547
- [Background] Steptoe A, Pollard TM, Wardle J. Development of a measure of the motives underlying the selection of food: the food choice questionnaire. Appetite. 1995 Dec;25(3):267-84. doi: 10.1006/appe.1995.0061. PMID 8746966
- [Background] Palombaro KM, Craik RL, Mangione KK, Tomlinson JD. Determining meaningful changes in gait speed after hip fracture. Phys Ther. 2006 Jun;86(6):809-16. PMID 16737406
- [Background] Whittaker JL, Emery CA. Sonographic measures of the gluteus medius, gluteus minimus, and vastus medialis muscles. J Orthop Sports Phys Ther. 2014 Aug;44(8):627-32. doi: 10.2519/jospt.2014.5315. Epub 2014 Jul 16. PMID 25029916
- [Background] Thomaes T, Thomis M, Onkelinx S, Coudyzer W, Cornelissen V, Vanhees L. Reliability and validity of the ultrasound technique to measure the rectus femoris muscle diameter in older CAD-patients. BMC Med Imaging. 2012 Apr 2;12:7. doi: 10.1186/1471-2342-12-7. PMID 22471726
- [Background] Schenkman M, Berger RA, Riley PO, Mann RW, Hodge WA. Whole-body movements during rising to standing from sitting. Phys Ther. 1990 Oct;70(10):638-48; discussion 648-51. doi: 10.1093/ptj/70.10.638. PMID 2217543
- [Background] Rosenberg JG, Ryan ED, Sobolewski EJ, Scharville MJ, Thompson BJ, King GE. Reliability of panoramic ultrasound imaging to simultaneously examine muscle size and quality of the medial gastrocnemius. Muscle Nerve. 2014 May;49(5):736-40. doi: 10.1002/mus.24061. PMID 24038069
- [Background] Pillen S, Tak RO, Zwarts MJ, Lammens MM, Verrijp KN, Arts IM, van der Laak JA, Hoogerbrugge PM, van Engelen BG, Verrips A. Skeletal muscle ultrasound: correlation between fibrous tissue and echo intensity. Ultrasound Med Biol. 2009 Mar;35(3):443-6. doi: 10.1016/j.ultrasmedbio.2008.09.016. Epub 2008 Dec 10. PMID 19081667
- [Background] Miyatani M, Kanehisa H, Ito M, Kawakami Y, Fukunaga T. The accuracy of volume estimates using ultrasound muscle thickness measurements in different muscle groups. Eur J Appl Physiol. 2004 Mar;91(2-3):264-72. doi: 10.1007/s00421-003-0974-4. Epub 2003 Oct 21. PMID 14569399
- [Background] Lindemann U, Muche R, Stuber M, Zijlstra W, Hauer K, Becker C. Coordination of strength exertion during the chair-rise movement in very old people. J Gerontol A Biol Sci Med Sci. 2007 Jun;62(6):636-40. doi: 10.1093/gerona/62.6.636. PMID 17595420
- [Background] Lindemann U, Claus H, Stuber M, Augat P, Muche R, Nikolaus T, Becker C. Measuring power during the sit-to-stand transfer. Eur J Appl Physiol. 2003 Jun;89(5):466-70. doi: 10.1007/s00421-003-0837-z. Epub 2003 Apr 24. PMID 12712354
- [Background] Fukumoto Y, Ikezoe T, Tateuchi H, Tsukagoshi R, Akiyama H, So K, Kuroda Y, Yoneyama T, Ichihashi N. Muscle mass and composition of the hip, thigh and abdominal muscles in women with and without hip osteoarthritis. Ultrasound Med Biol. 2012 Sep;38(9):1540-5. doi: 10.1016/j.ultrasmedbio.2012.04.016. Epub 2012 Jun 30. PMID 22749818
- [Derived] Ryan AS, Beamer BA, Gruber-Baldini AL, Craik RL, Golden J, Guralnik J, Hochberg MC, Mangione KK, Orwig D, Rathbun AM, Magaziner J. Effects of Multicomponent Home-Based Intervention on Muscle Composition, Fitness, and Bone Density After Hip Fracture. J Gerontol A Biol Sci Med Sci. 2024 May 1;79(5):glae078. doi: 10.1093/gerona/glae078. PMID 38452133
- [Derived] Huang MZ, Rogers MW, Pizac D, Gruber-Baldini AL, Orwig D, Hochberg MC, Beamer BA, Creath RA, Savin DN, Conroy VM, Mangione KK, Craik R, Zhang LQ, Magaziner J. Effect of Multicomponent Home-Based Training on Gait and Muscle Strength in Older Adults After Hip Fracture Surgery: A Single Site Randomized Trial. Arch Phys Med Rehabil. 2023 Feb;104(2):169-178. doi: 10.1016/j.apmr.2022.08.974. Epub 2022 Sep 7. PMID 36087806
- [Derived] Mutchie HL, Orwig DL, Beamer B, Conroy V, Guralnik J, Magaziner J, Gruber-Baldini AL. Four Square Step Test Performance in Hip Fracture Patients. J Geriatr Phys Ther. 2022 Apr-Jun 01;45(2):81-89. doi: 10.1519/JPT.0000000000000310. PMID 33935219
- [Derived] Magaziner J, Mangione KK, Orwig D, Baumgarten M, Magder L, Terrin M, Fortinsky RH, Gruber-Baldini AL, Beamer BA, Tosteson ANA, Kenny AM, Shardell M, Binder EF, Koval K, Resnick B, Miller R, Forman S, McBride R, Craik RL. Effect of a Multicomponent Home-Based Physical Therapy Intervention on Ambulation After Hip Fracture in Older Adults: The CAP Randomized Clinical Trial. JAMA. 2019 Sep 10;322(10):946-956. doi: 10.1001/jama.2019.12964. PMID 31503309
- [Derived] Orwig D, Mangione KK, Baumgarten M, Terrin M, Fortinsky R, Kenny AM, Gruber-Baldini AL, Beamer B, Tosteson A, Shardell M, Magder L, Binder E, Koval K, Resnick B, Craik RL, Magaziner J. Improving community ambulation after hip fracture: protocol for a randomised, controlled trial. J Physiother. 2017 Jan;63(1):45-46. doi: 10.1016/j.jphys.2016.10.001. Epub 2016 Oct 28. PMID 27964962

DOCUMENTS (2):
  • Study Protocol (2016-10-19): https://cdn.clinicaltrials.gov/large-docs/04/NCT01783704/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-01): https://cdn.clinicaltrials.gov/large-docs/04/NCT01783704/SAP_002.pdf